CLINICAL TRIAL: NCT00340665
Title: Study of Estrogen Activity & Development (SEAD) SEAD2: Physical Exam and Ballard Markers; Sead 3: Biochemistry
Brief Title: Study of Infant Diets on Estrogen Activity and Development
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999903184; 03-E-N184
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2019-11-21 (Actual); Status verified 2012-08-22

CONDITIONS: Infant Formula; Estrogen Activity
Keywords: Soy; Infant Formula; Sexual Development; Hormone; Isoflavones

SUMMARY:
This study, conducted at the University of Pennsylvania s Newborn Nursery, the Children s Hospital of Philadelphia, and the Exton Specialty Care Center, will examine how different infant diets may affect estrogen activity in babies. During pregnancy, babies are exposed to the female hormone estrogen from their mother. Estrogen plays a key role in the development of breasts and milk production, as well as the development of the uterus. The effects of these hormones can be seen when babies are examined. Between 6 and 12 months of age, the effects are reduced. Breast milk and some infant formulas may contain compounds that can act like female hormones in the body and may prolong the estrogen effects.

This study has two parts. Part 1 studies the physical development of babies fed different ways. Part 2 studies how hormone levels in babies differ depending on what they are being fed. Babies may participate in one or both parts. Part 1 includes babies 0 to 6 months of age; part 2 includes babies 0 to 12 months of age. In each part of the study, parents may choose to have their babies evaluated from one to four times.

Full-term infants (age 37 to 41 weeks gestational age) from birth to 12 months of age who weigh from 2501 to 4499 grams (about 5.5 to 10 pounds) at birth and who have no chromosomal abnormalities, major malformations, or endocrine problems may be eligible for this study. Male infants must have palpable testes. Infants being fed a diet of breast milk, soy milk, or cow s milk will be included. Study procedures include the following:

Part 1

* Feeding history: the parent provides information about the baby s dietary intake since birth.
* Length, weight, and head circumference: the baby s measurements are taken.
* Physical examination: the baby s physical maturity is assessed by examination of the skin, breasts, and external sex organs.
* Breast secretions: the baby s breast buds are gently pressed during the physical examination to look for a milky-white substance that some babies produce during the first year of life. If the substance appears, a specimen will be collected.
* Vaginal cells: for baby girls, the opening of the vaginal area is gently swabbed with a sterile Q-tip to assess the maturity of the vaginal lining.

Part 2

* Feeding history and length, weight and head circumference measurements as described above.
* Urine: a urine sample is collected in a cotton diaper or a urine collection bag.
* aliva: a saliva sample is collected by gently swabbing the inside of the baby s mouth 1 hour after a morning feeding to remove any left over milk.
* Hair: a lock of hair, 1/2-inch wide and 1 to 2 inches long is taken from 12-month old babies.
* Blood: some infants have a small blood sample collected by a heel-stick.

This study will serve as a basis for a later study about how infant formulas affect infant growth.

DETAILED DESCRIPTION:
Term newborns have anatomic and sonographic evidence of in utero estrogen exposure. Over the first six months to a year of life, as the influence of maternal hormone wanes, these findings recede. Soy infant formula contains large amounts of isoflavones (diadzein and genistein) that can occupy estrogen receptors and act as estrogens in the laboratory. A food substance with estrogen activity might prolong the effect of maternal hormones, or interfere with hormonal homeostasis the child. Two cross-sectional pilot study (SEAD 2 and SEAD 3) will be undertaken in order to establish the methods for a future, multi-center study designed to assess the potential effects of soy formula on estrogen activity in infants. Another cross-sectional pilot study (SEAD 1) will be undertaken to evaluate anatomical evidence detected by ultrasound and will be conducted at The Children's Hospital in Boston. Details of the SEAD 1 study will not be presented in this protocol. In the first pilot study (SEAD 2), 84 examinations of full-term infants, ages 0-6 months and on one of three feeding regimens (soy formula, breast milk or cow's milk formula) will be conducted. This study will establish a protocol for examining and sampling methods to be used for a later trial investigating whether exposure to soy estrogen compared to breast milk and non-soy formulas prolongs anatomical evidence of estrogen exposure and response. In addition to the physical examination, vaginal cells will be collected for cytology analysis. Breast nipple secretions, if present, will also be collected and analyzed for protein and sugar levels. In the second pilot study (SEAD 3), 372 evaluations on full-term infants will be conducted in parallel with the first study. SEAD 3 will assess the hormonal and biochemical status of full-term infants age 0-12 months. This study will establish a protocol for sampling methods to be used for collecting urine, saliva, serum, and hair samples. Endogenous hormone levels such as testosterone, estradiol, and isoflavone levels (genestein and diadzein) will be measured in serum and the results will be compared against the non-serum tests (urine, saliva and hair). The purpose of these two pilot studies is twofold. The first is to develop and finalize recruitment and collections procedures in preparation for a larger, comprehensive trial of biological response in children to soy formula with and without the estrogenic isoflavones. The second is to study the natural history of estrogen activity in infants on a variety of feeding regimens.

ELIGIBILITY:
* INCLUSION CRITERIA:

SEAD 2 and 3

1. Full term infants defined as age 37-41 weeks gestational age at birth. Ultrasound evidence or reliable reporting of last menstrual period (LMP) by infant's mother.
2. Can be categorized into one of the feeding definitions.
3. Birth weight between 2501-4499 grams.
4. Age 0-6 months for SEAD 2, age 0-12 months for SEAD 3
5. For SEAD 3, for 12-months age interval, subjects must not have had first haircut.

EXCLUSION CRITERIA:

SEAD 2 and 3

1. Chromosomal aberrations
2. Major malformation
3. SEAD 2: Non-palpable testis (males only)
4. Presence of an endocrinopathy (i.e., ambiguous genitalia, congenital hypothyroidism)

This is a natural history study and children must be healthy in order to participate in this study. Therefore, children will be excluded from the study if they are known to have chromosomal aberrations, or any major malformations or an endocrinopathy. Testicular development is an important endpoint in this study and therefore males will be excluded from SEAD 2 if the testes are not palpable.

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 239 (Actual)
Dates: Start 2003-05-05; Study Completion 2012-08-22

CONTACTS AND LOCATIONS:
Overall Officials: Walter Rogan, M.D., Principal Investigator — National Institute of Environmental Health Sciences (NIEHS)
Locations (2):
- United States (2):
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Childrens Hospital, Philadelphia, Philadelphia, Pennsylvania

REFERENCES:
- [Background] Setchell KD, Zimmer-Nechemias L, Cai J, Heubi JE. Isoflavone content of infant formulas and the metabolic fate of these phytoestrogens in early life. Am J Clin Nutr. 1998 Dec;68(6 Suppl):1453S-1461S. doi: 10.1093/ajcn/68.6.1453S. PMID 9848516
- [Background] Cruz ML, Wong WW, Mimouni F, Hachey DL, Setchell KD, Klein PD, Tsang RC. Effects of infant nutrition on cholesterol synthesis rates. Pediatr Res. 1994 Feb;35(2):135-40. doi: 10.1203/00006450-199402000-00001. PMID 8165045
- [Background] Strom BL, Schinnar R, Ziegler EE, Barnhart KT, Sammel MD, Macones GA, Stallings VA, Drulis JM, Nelson SE, Hanson SA. Exposure to soy-based formula in infancy and endocrinological and reproductive outcomes in young adulthood. JAMA. 2001 Aug 15;286(7):807-14. doi: 10.1001/jama.286.7.807. PMID 11497534